CLINICAL TRIAL: NCT04949724
Title: Psychometric Properties of The Turkish Health Enhancement Lifestyle Profile-Screener Questionnaire (T-Help-Screener)
Brief Title: Turkish Health Enhancement Lifestyle Profile-Screener Questionnaire
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İnal, principal investigator, Trakya University
Other Study IDs: 2018/101
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Elderly Population
MeSH Terms: interventions — Protein Biosynthesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: translation and adaptation study — translation and adaptation study

SUMMARY:
The aim of this study was to evaluate the validity, reliability, and cultural adaptation of the Turkish version of the Health Enhancement Lifestyle Profile Screener (T-HELP-Screener).

DETAILED DESCRIPTION:
Internal consistency of the T-HELP-Screener was measured using Kuder-Richardson. Test-retest reliability was performed with 66 of the 150 participants using intraclass correlation coefficient (ICC). Construct validity of the T-HELP-Screener was analyzed with the Healthy Lifestyle Behavior Scale-II (HLBS-II).

ELIGIBILITY:
Inclusion Criteria:

age over 65 years, no communication problems, and a Mini-Mental State Examination score of 24 or above

Exclusion Criteria:

communication problem

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: elderly people
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Behavior Scale-II | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Özgü İnal, Ankara, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No